CLINICAL TRIAL: NCT00547638
Title: Multicenter, Prospective, Randomized Controlled Study to Show Equivalence of DERMABOND PROTAPE to DERMABOND HVD for Closure of Simple, Thoroughly Cleansed, Trauma-induced Wounds in the Emergency Department
Brief Title: Study to Show Equivalence of DERMABOND PROTAPE to DERMABOND HVD for Wound Closure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07CS005; IDE Number:G060268 (Other: FDA)
Record Dates: First submitted 2007-10-17; First posted 2007-10-22 (Estimated); Results first posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Lacerations
Keywords: laceration/wound closure; topical skin adhesive
MeSH Terms: conditions — Lacerations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dermabond Protape (Experimental): DERMABOND PROTAPE (Prineo) Topical Skin Adhesive
  Interventions: Device: cyanoacrylate with pressure sensitive mesh
- Dermabond HVD (Active Comparator): DERMABOND HVD Topical Skin Adhesive
  Interventions: Device: cyanoacrylate

INTERVENTIONS:
Device: cyanoacrylate with pressure sensitive mesh — Topical Skin Adhesive
  Other Names: Dermabond Protape; Prineo
  Arms: Dermabond Protape
Device: cyanoacrylate — Topical Skin Adhesive
  Other Names: Dermabond - HVD; Dermabond - Protape
  Arms: Dermabond HVD

SUMMARY:
This is a multicenter, prospective, randomized controlled study for the purpose of comparing DERMABOND PROTAPE to DERMABOND HVD for closure of wounds in the Emergency Department. The objective of this study is to demonstrate whether the incidence of wound closure for DERMABOND PROTAPE is equivalent to that measured for DERMABOND HVD.

DETAILED DESCRIPTION:
According to the literature, cyanoacrylate adhesives (topical skin adhesive) have performed as intended and have not produced results that would bring into question the safety or effectiveness of cyanoacrylate adhesive for closure of surgical incisions and traumatic wounds in humans.

As such, this is a multicenter, prospective, randomized controlled study for the purpose of comparing two forms of topical skin adhesives, DERMABOND PROTAPE & DERMABOND HVD for closure of wounds in the Emergency Department.

Patients presenting in the Emergency Department with traumatic wounds meeting the acceptance criteria will have their wounds closed with DERMABOND PROTAPE or DERMABOND HVD, and will be monitored and evaluated at 14 & 30 days.

ELIGIBILITY:
Inclusion Criteria:

* at least 1 year of age
* in good general health in the opinion of the Investigator.
* have at least one traumatic wound meeting the criteria for closure as defined in current Dermabond product labeling.
* patient must be willing to follow instructions for wound care listed in device labeling and refrain from picking at the device, applying topical medications to the wound, and swimming or soaking in a tub until the sutures are removed.
* patient agrees to return for follow-up evaluation
* patient (or guardian) signs the informed consent
* patient is reasonably expected to survive the study

Exclusion Criteria:

* significant multiple trauma (merely multiple wounds are allowed)
* peripheral vascular disease
* insulin dependent diabetes mellitus
* known to have a blood clotting disorder
* receiving antibiotic therapy for preexisting condition or infection
* known to be HIV-positive or otherwise immunocompromised
* known personal or family history of keloid formation or hypertrophy
* currently taking systemic steroids
* known allergy to cyanoacrylate, formaldehyde, tapes or adhesives
* participating in another current clinical study
* history of abnormal wound healing
* burst stellate lacerations due to a crush or hard blow
* animal or human bite or scratch
* decubitus ulcer
* puncture wound
* wound at mucocutaneous junction or in mucosal (but not excluding the vermillion border of the lip)
* wound on scalp covered by natural hair
* wound has visual evidence of active infection
* gangrenous wound
* wound requiring debridement of devitalized or contaminated tissue
* wound at site of active rash/skin lesion making evaluation difficult
* previously treated wound or has failed to heal
* wound in high skin tension area or across an area of increased skin tension, such as knuckles, elbows, or knees, unless the joint will be immobilized during the skin healing period or unless skin tension has been removed by application

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2007-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Colquhoun, MD, Study Director — Pleiad Devices
Locations (9):
- United States (9):
  - NextCare Institute For Clinical Research, Phoenix, Arizona
  - Orlando Regional Healthcare System, Orlando, Florida
  - Investigators Research Group, LLC, Indianapolis, Indiana
  - Tulane Universtiy Hospital & Clinic, New Orleans, Louisiana
  - Stony Brook University HSC, Stony Brook, New York
  - Duke University Health System, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Drexel University Hospital, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects were recruited from the general population ≥1 year of age who were treated in an Emergency Department/Urgent Care Setting.
Groups:
- Dermabond Protape (Prineo): DERMABOND PROTAPE (Prineo: Tissue adhesive for topical application.
- Dermabond HVD: DERMABOND HVD: Comparator tissue adhesive for topical application.
Period: Overall Study
Arm/Group | Dermabond Protape (Prineo) | Dermabond HVD
Started | 143 | 73
Completed | 119 | 59
Not Completed | 24 | 14

BASELINE CHARACTERISTICS:
Groups:
- Dermabond Protape (Prineo): DERMABOND PROTAPE (Prineo) Tissue adhesive for Topical Application
- Total: Total of all reporting groups
Arm/Group | Dermabond Protape (Prineo) | Dermabond HVD | Total
Number analyzed (Participants) | 143 | 73 | 216
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 52 | 30 | 82
  Between 18 and 65 years | 89 | 39 | 128
  >=65 years | 2 | 4 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 25.0 (18.4) | 25.7 (19.8) | 25.2 (18.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 26 | 78
  Male | 91 | 47 | 138
Region of Enrollment [Number; unit: Participants]
  United States | 143 | 73 | 216

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of Wound Closure Post-treatment, as Defined by Continuous Approximation of Wound Margins From the Time of Wound Closure Until the Day of Evaluation Without Dehiscence or Need for Reclosure.
Description: Data is presented as binomial tables of proportions of successes and failures for each treatment. The 90% two-sided exact confidence intervals (CI) for the differences in the proportions for each study group was calculated. The upper limit of the 90% CI was then taken to represent the upper limit of the one-sided 95% CI. The primary objective of the study was met if the upper limit of the one-sided 95% CI of the difference in proportions (comparator minus treatment) did not exceed 8%.
Time Frame: 14 days (±2 days)
Population: Intent to treat population results are presented.With respect to Measure Description it is defined as the number of participants in each group with successful wound-closure (approximation).
Measure: Number; unit: Participants
Arm/Group | Dermabond Protape (Prineo) | Dermabond HVD
Number analyzed (Participants) | 143 | 73
Participants | 123 | 57
Statistical Analysis 1: Comparison: Dermabond Protape (Prineo) vs Dermabond HVD; Test type: Non-Inferiority or Equivalence — Equivalence is demonstrated if the upper limit of the 95% confidence interval (when subtracting the percentage of DERMABOND PROTAPE successful subjects from the percentage of DERMABOND HVD successful subjects) does not exceed 8%; Gart-Nam; Difference in Proportion of Successes = -7.9, 95% CI 2-sided [-17.7 to 1.0] — The value for the Estimated Parameter is expressed as a percentage and is defined as the difference in the proportion of sucesses between study groups

2. Secondary Outcome: Cosmesis
Description: The evaluation of healing and cosmetic outcome post-treatment using the modified Hollander Cosmesis Scale (mHCS). The proportion of patients with a zero (0) score will be compared between the test and control arms.
Time Frame: 30 days (±5 days)
Population: Intent to Treat Population where good outcome for overall appearance. A p-value of 0.457 was determined following comparison by Fisher's Exact Test.
Measure: Number; unit: Participants
Arm/Group | Dermabond Protape (Prineo) | Dermabond HVD
Number analyzed (Participants) | 143 | 73
Participants | 93 | 43
Statistical Analysis 1: Comparison: Dermabond Protape (Prineo) vs Dermabond HVD; Test type: Superiority or Other; p = 0.457, Fisher Exact — The total mHCS scores are summarized as proportion of subjects with good outcome (total scores of zero) and a comparison of treatment groups by Fisher Exact Test was performed to confirm differences in groups

3. Other Pre Specified Outcome: The Comparison of Test and Control Arms Regarding Incidence of Clinical Infection at Day 14 and Day 30
Description: Incidence of clinical infection (defined by observation of redness, swelling, purulent discharge, pain, increased skin temperature, fever or other systemic signs of injection) collected at the Day 14 and Day 30 visits. A formal statistical analysing using Fisher's Exact Test was performed.
Time Frame: Through Day 30
Population: Intent to treat population was analyzed for the presence of signs of infection at Day 14 and Day 30.
Measure: Number; unit: Participants
Arm/Group | Dermabond Protape (Prineo) | Dermabond HVD
Number analyzed (Participants) | 143 | 73
Participants
  Number of Infections at Day 14 Per Group | 4 | 1
  Number of Infections at Day 30 Per group | 2 | 0
Statistical Analysis 1: Comparison: Dermabond Protape (Prineo) vs Dermabond HVD; Test type: Superiority or Other; p = 1.0000, Fisher Exact — Differences between treatment groups in the incidence rate of infection at Day 14 and Day 30 were compared using the Fisher's Exact Test
Statistical Analysis 2: Comparison: Dermabond Protape (Prineo) vs Dermabond HVD; Test type: Superiority or Other; p = 1.0000, Fisher Exact — Differences between treatment groups in the incidence rate of infection at Day 30 were compared using the Fisher's Exact Test

4. Other Pre Specified Outcome: The Incidence and Extent of Local Acute Inflammatory Reactions Including Edema, Erythema, Pain and Local Temperature at Day 14 and Day 30
Description: Each parameter (edema, erythema, pain and location temperature) is measured on a 4 point scale (0, 1, 2, 3). The individual values are added to generate an overall AIRE Score. AIRE Scores were summarized as good (score=0) versus poor (score>0) by treatment group and compared for differences using the Fisher's Exact Test.
Time Frame: At Day 14 and Day 30
Population: Intent to treat population was analyzed for subjects in each group with Total AIRE Score of 1-12 at Day 14 and Day 30. Analysis is performed on the proportion of subjects in each group with Total AIRE Scores greater than 0 versus those less or equal to 0 at each timepoint.
Measure: Number; unit: Participants With AIRE Score >0
Arm/Group | Dermabond Protape (Prineo) | Dermabond HVD
Number analyzed (Participants) | 143 | 73
Participants With AIRE Score >0
  Participants with Total AIRE Score >0 at Day 14 | 54 | 35
  Participants with Total AIRE Score >0 at Day 30 | 55 | 29
Statistical Analysis 1: Comparison: Dermabond Protape (Prineo) vs Dermabond HVD; Test type: Superiority or Other; p = 0.188, Fisher Exact — Intent to treat population was analyzed
Statistical Analysis 2: Comparison: Dermabond Protape (Prineo) vs Dermabond HVD; Test type: Superiority or Other; p = 0.883, Fisher Exact — Intent to treat population was analyzed

5. Other Pre Specified Outcome: Incidence of Skin Blistering at Day 14
Description: The incidence of skin blistering is presented as a tabulation of the presence or absence of skin blistering by treatment group. A formal statistical analysis of the incidence of blistering at Day 14 was performed using the Fisher's Exact Test.
Time Frame: Day 14
Population: Intent to treatment population was analyzed for the incidence of skin blistering at Day 14.
Measure: Number; unit: Participants With Blistering at Day 14
Arm/Group | Dermabond Protape (Prineo) | Dermabond HVD
Number analyzed (Participants) | 143 | 73
Participants With Blistering at Day 14 | 0 | 0
Statistical Analysis 1: Comparison: Dermabond Protape (Prineo) vs Dermabond HVD; Test type: Superiority or Other; p = 1.0000, Fisher Exact

6. Other Pre Specified Outcome: Incidence of Any Other Anticipated or Unanticipated Adverse Events
Description: Adverse events were coded using the MedDRA dictionary. In addition severity, relationship to treatment and procedure, action taken and outcome were described. Adverse events were summarized by treatment group. No formal statistical analysis was performed on overall incidence of adverse events with the exception of clinical infection, acute inflammatory reactions and skin blistering.
Time Frame: Day 30
Population: Intent to treat population in which subjects experiencing at least 1 adverse event were reported and analyzed.
Measure: Number; unit: Participants Experiencing at least 1 AE
Arm/Group | Dermabond Protape (Prineo) | Dermabond HVD
Number analyzed (Participants) | 143 | 73
Participants Experiencing at least 1 AE | 34 | 10

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from time of treatment out through Day 30.
Description: The incidence of adverse events were compared between treatment groups.
Arm/Group | Dermabond Protape (Prineo) | Dermabond HVD
Serious Adverse Events (participants affected / at risk) | 0/143 | 0/73
Other Adverse Events (participants affected / at risk) | 0/143 | 0/73

LIMITATIONS AND CAVEATS:
The percentages of participants who withdrew prematurely from the study from each group could represent a possible study limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less